CLINICAL TRIAL: NCT00317174
Title: Assess Immune Persistence & Memory by Giving Plain PRP,PSA & PSC (10 Mths Age), & Immunogenicity & Safety of a Tritanrix™-HBV/Hib-MenAC/ Tritanrix™-HBV/Hib2.5 Booster (15-18 Mths Age) in Previously Primed Subjects
Brief Title: A Study to Assess Antibody Persistence, Boostability & Safety in Previously Primed Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 759346/002
Record Dates: First submitted 2006-02-15; First posted 2006-04-24 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b; Tetanus; Whole Cell Pertussis; Hepatitis B; Diphtheria
MeSH Terms: conditions — Haemophilus Infections; Tetanus; Hepatitis B; Diphtheria

INTERVENTIONS:
Biological: DTPw-HBV/Hib-MenAC conjugate vaccine

SUMMARY:
The purpose of the study is as follows:

* To evaluate the persistence of antibodies and the presence of immune memory induced by a 3-dose primary vaccination with Tritanrix™-HepB/Hib-MenAC (three formulations) in the study DTPwHB/HibMenACTT001 (CPMS No. 759346/001) by giving unconjugated PRP, PSA and PSC at 10 months age to one subset of subjects.
* To evaluate the persistence of all antibodies pertaining to primary vaccination and the booster response to Tritanrix™-HepB/Hib2.5 vaccine or Tritanrix™-HepB/Hib-MenAC vaccine at 15-18 months age in the other subset of subjects.

DETAILED DESCRIPTION:
This study will be conducted in two stages:

At 10 months age, half of the subjects will receive a dose of plain meningococcal AC and PRP polysaccharide (PS) vaccine at 10 months age.

At 15 to 18 months age (DTP booster phase), all subjects will receive a booster dose of Tritanrix™-HepB/Hib-MenAC or Tritanrix™-HepB/Hib2.5.

ELIGIBILITY:
Inclusion criteria:

• Healthy child 10 months that participated in the study DTPwHB/HibMenACTT001 (CPMS No. 759346/001), written informed consent obtained from the parents.

Exclusion criteria:

* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before and ending 30 days after administration of study vaccines with the exception of oral polio vaccine (OPV).
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during study period.
* Chronic administration (> 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Previous booster vaccination against diphtheria, tetanus, pertussis, hepatitis B, serogroups A or C meningococcal disease and/or Hib since the last visit of study 759346/001.
* History of/known exposure to diphtheria, tetanus, pertussis, hepatitis B, serogroups A or C meningococcal and/or Hib disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.

Min Age: 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450
Dates: Start 2003-07; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Pre & 1M post-plain PS, antibody levels & bactericidal titers (meningococcal serogroups A & C). Pre & 1M post-DTP booster, antibody levels for all vaccine antigens.

SECONDARY OUTCOMES:
Pre & 1M post-DTP booster (subset of subjects), antibody levels for all vaccine antigens. Retrospective serious adverse events (SAEs). Solicited (day 0-7), unsolicited events (day 0-30). SAEs (entire study)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gatchalian S, Palestroque E, De Vleeschauwer I, Han HH, Poolman J, Schuerman L, Dobbelaere K, Boutriau D. The development of a new heptavalent diphtheria-tetanus-whole cell pertussis-hepatitis B-Haemophilus influenzae type b-Neisseria meningitidis serogroups A and C vaccine: a randomized dose-ranging trial of the conjugate vaccine components. Int J Infect Dis. 2008 May;12(3):278-88. doi: 10.1016/j.ijid.2007.08.007. Epub 2007 Nov 5. PMID 17981067
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 759346/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 759346/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 759346/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 759346/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 759346/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 759346/002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register